CLINICAL TRIAL: NCT03148210
Title: A Randomized, Controlled, Clinical Trial to Address the Burden of Undiagnosed Airflow Obstruction in Canadian Adults
Brief Title: Undiagnosed COPD and Asthma Population Study (UCAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20170182-01H
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Care (Active Comparator): Treatment strategy using evidence-based guidelines for asthma or COPD
  Interventions: Drug: Treatment strategy using evidence-based guidelines for asthma or COPD; Behavioral: Smoking Cessation; Behavioral: Participant Education
- Standard of Care (Placebo Comparator): Spirometry result sent to family MD
  Interventions: Behavioral: Smoking Cessation

INTERVENTIONS:
Drug: Treatment strategy using evidence-based guidelines for asthma or COPD — The respirologist will determine the clinical extent of the patient's symptoms, activity limitation, and degree of airflow obstruction and will commence the subject on asthma or COPD medications if indicated
  Arms: Enhanced Care
Behavioral: Smoking Cessation — Smoking cessation counselling by a qualified educator if currently smoking
Behavioral: Participant Education — Standardized education for asthma or COPD disease
  Arms: Enhanced Care

SUMMARY:
Previous population health studies suggest that up to 10% of Canadian adults have undiagnosed asthma or COPD- these people are currently undiagnosed and untreated, even though they may have significant respiratory symptoms. Our study will use targeted casefinding to find people with undiagnosed asthma and COPD in Canadian communities. The investigators will assess their symptoms and their health care use and number of sick days to determine the burden of undiagnosed respiratory disease in these people. The investigators will then determine whether early treatment of previously undiagnosed airflow obstruction will improve patients' health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 18 years old;
* Subjects who score > or = to 6 points on The Asthma Screening Questionnaire or > 19.5 points on The COPD Diagnostic Questionnaire;
* Subjects who have given written informed consent to participate in this trial in accordance with local regulations;
* Subjects able to perform pre and post bronchodilator spirometry to measure lung function;

Additional Inclusion Criteria for RCT:

Those subjects who have undiagnosed airflow obstruction (i.e. Asthma will be diagnosed in subjects with airflow obstruction whose FEV1 improves by > 12% and 200 ml after bronchodilator and COPD will be diagnosed in subjects who do not have a significant bronchodilator response and who exhibit persistent airflow obstruction post bronchodilator) will be asked to consent and participate in the RCT.

Exclusion Criteria:

* Subjects who report a previous physician diagnosis of asthma.
* Subjects who report a previous physician diagnosis of COPD
* Subjects with any of the following conditions within the past 3 months: Heart attack or hospitalization for other heart problems; Stroke; Aortic or cerebral aneurysm; Detached retina or eye surgery
* Subjects who are in the third trimester of pregnancy
* Subjects involved in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Annual rate of patient initiated healthcare utilization events for respiratory illness | 12 months
  Number of visits for respiratory illnesses divided by the length of time in the study

SECONDARY OUTCOMES:
Changes in forced expiratory volume in one second (FEV1) measured in litres (L) using pre bronchodilator spirometry testing and post bronchodilator spirometry testing. | 12 months
  The change will be expressed as the mean change in the FEV1 measurements at 12 months in comparison to the lung function measurements on the day of randomization.
Quality of life changes as assessed by the 36-Item Short Form Health Survey (SF-36) Health Survey Questionnaire | 12 months
  The change in general health status will be expressed as the total score of the SF-36 Health Survey Questionnaire at 12 months minus the score on the day of randomization. A total change of 8-10 points in the SF-36 has been established as the minimal clinically important difference (MCID) for this questionnaire. Higher scores indicate better health status.
Change in disease-specific quality of life quantified using the St. George's Respiratory Questionnaire (SGRQ). | 12 months
  The change in disease-specific quality of life will be expressed as the total St. George's Respiratory Questionnaire score at 12 months minus the score on the day of randomization. This questionnaire includes 3 domains: symptoms (distress caused by specific respiratory symptoms); activity (physical activities that cause or are limited by breathlessness); and impact (social and psychological effects of the respiratory disease). A total change of - 4 points in the SGRQ total score has been established as the minimal clinically important difference (MCID) for this questionnaire. Higher scores indicate poor health status.
Changes in overall respiratory symptoms (including cough, sputum and dyspnea) will be assessed using the COPD Assessment Test (CAT) | 12 months
  The change in overall respiratory symptom burden will be expressed as the total score of the COPD Assessment Test at 12 months minus the score on the day of randomization. A total change of - 2 points in the CAT total score has been established as the minimal clinically important difference (MCID) for this questionnaire. Higher scores indicate higher burden.
Smoking cessation rate | 12 months
  The number of participants who quit smoking over the 12 month period.

CONTACTS AND LOCATIONS:
Locations (15):
- Canada (15):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital- The Lung Centre, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - St. Clare's Mercy Hospital, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Firestone Institute for Respiratory Health, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital-General Campus, Ottawa, Ontario
  - St. Micheal's Hospital, Toronto, Ontario
  - The Research Institute of the McGill University Health Centre (RI-MUHC), Montreal, Quebec
  - Hopital du Scaré-Coeur, Montreal, Quebec
  - IUCP, Hôpital Laval, Québec, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aaron SD, Vandemheen KL, Whitmore GA, Bergeron C, Boulet LP, Cote A, McIvor RA, Penz E, Field SK, Lemiere C, Mayers I, Bhutani M, Azher T, Lougheed MD, Gupta S, Ezer N, Licskai CJ, Hernandez P, Ainslie M, Alvarez GG, Mulpuru S; UCAP Investigators. Early Diagnosis and Treatment of COPD and Asthma - A Randomized, Controlled Trial. N Engl J Med. 2024 Jun 13;390(22):2061-2073. doi: 10.1056/NEJMoa2401389. Epub 2024 May 19. PMID 38767248